CLINICAL TRIAL: NCT05478590
Title: HR POSITIVE, HER 2 NEGATIVE ADVANCED BREAST CANCER- TREATMENT PATTERNS IN POLAND - HABER STUDY
Brief Title: A Study to Describe Treatment Patterns of Advanced Breast Cancer in Poland in the Real-world Data Setting
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5481177
Record Dates: First submitted 2022-07-26; First posted 2022-07-28 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Breast Neoplasms
Keywords: Hormone receptor-positive human epidermal growth factor receptor 2 negative (HR+ HER2-); advanced breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
The study is descriptive and aims to characterize the treatment patterns of advanced breast cancer in Poland in the real-world data setting. The main goals are to assess the current treatment patterns of hormone receptor-positive (HR+) Human epidermal growth factor receptor 2 negative (HER2-) advanced breast cancer and their changes in clinical practice and relate them to patients' demographics, disease characteristics, type of other therapies used in patients as well as disease progression and visceral crisis occurrence.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with histologically diagnosed advanced breast cancer (with locoregional recurrence not eligible for radical local treatment or with distant metastases)
* Patient has a documented hormone (estrogen and/or progesterone) receptor expression and lack of HER2 receptor overexpression or lack of HER2 gene amplification (HR+/HER2- breast cancer subtype)
* Patient had no prior treatment for advanced breast cancer
* Patient has no symptomatic metastases to the central nervous system
* There is no other malignancies in patient requiring active treatment
* Patient is without co-occurring other malignancies treated with palliative assumption

Exclusion Criteria:

* Parallel patient's participation in any other clinical trial at the time when the decision over the advanced breast cancer treatment was made or up to 30 days before it.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients treated for the locally advanced/metastatic breast cancer of the HR+ HER2- subtype
Sampling Method: Non-Probability Sample
Enrollment: 440 (Actual)
Dates: Start 2021-11-22 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants With HR+ HER2- Advanced Breast Cancer (ABC) Treatment Patterns | 01 September 2020 through 31 August 2021

SECONDARY OUTCOMES:
Number of Changes in Clinical Practice During One Year Observational Period in Relation to the Local Breast Cancer (BC) Treatment Guidelines | 01 September 2020 through 31 August 2021
Correlation of Treatment Patterns With the Reference of the si.+-te Defined by Number of Enrolled Patients | 01 September 2020 through 31 August 2021
Demographical Characteristics of Participants | 01 September 2020 through 31 August 2021
Correlation of Treatment Type to Demographical Characteristics of Participants | 01 September 2020 through 31 August 2021
Disease Characteristics of Treated BC Participants | 01 September 2020 through 31 August 2021
Clinical Characteristics of Treated BC Participants | 01 September 2020 through 31 August 2021
Treatment Modalities of Neoadjuvant Therapies Early BC | 01 September 2020 through 31 August 2021
  In this outcome measure participants with different treatment modalities including hormonotherapy and chemotherapy
Treatment Modalities of Adjuvant Therapies Early BC | 01 September 2020 through 31 August 2021
  In this outcome measure participants with different treatment modalities including hormonotherapy and chemotherapy
Time to Disease Free Interval | 01 September 2020 through 31 August 2021
  Last Dose of Last Drug Taken in Adjuvant Treatment
Number of Participants With Association Between Disease Characteristic and ABC Treatment Patterns | 01 September 2020 through 31 August 2021
Number of Participants With Association Between Clinical Characteristic and ABC Treatment Patterns | 01 September 2020 through 31 August 2021
Number of Participants With Association Between Neoadjuvant Therapy and ABC Treatment Patterns | 01 September 2020 through 31 August 2021
Number of Participants With Association Between Adjuvant Therapy and ABC Treatment Patterns | 01 September 2020 through 31 August 2021
Number of Participants With Association Between Time to Relapse in early BC Treatment and ABC Treatment Patterns | 01 September 2020 through 31 August 2021
Number of Participants With Association Between Concomitant Therapy and ABC Treatment Patterns | 01 September 2020 through 31 August 2021
Proportion of Participants With Diagnosed Visceral Crisis | 01 September 2020 through 31 August 2021
Number of Visceral Crisis Diagnosis in Compliance With ABC5 Guidelines | 01 September 2020 through 31 August 2021
  ABC5 guideline definition visceral crisis (updated in 2020) is a severe organ disfunction that involve: Severe symptoms and signs, rapid disease progression, and laboratory values

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (19):
- Poland (19):
  - Ambulatorium Chemioterapii Centrum Onkologii, Bydgoszcz
  - Wojewodzki Szpital Zespolony w Elblągu - oddzial onkologii, Elblag
  - Uniwersyteckie Centrum Kliniczne, Klinika Onkologii i Radioterapii, Gdansk
  - Oddział onkologii Szpital Specjalistyczny im. H. Klimontowicza, Gorlice
  - Oddział Onkologii Klinicznej, Kalisz
  - Narodowy Instytut Onkologii, Krakow
  - Oddział Onkologii Klinicznej z Pododdziałem Dziennym, Krakow
  - Klinika Onkologii, Instytut Centrum Zdrowia Matki Polki, Lodz
  - Opolskie Centrum Onkologii, Opole
  - Oddział/Poradnia Onkologiczna Wojewodzki Szpital w Przemyślu, Przemyśl
  - Podkarpackie Centrum Onkologii, Rzeszów
  - SPZOZ Oddział onkologii klinicznej, Swidnica
  - Zachodniopomorskie Centrum Onkologii, Szczecin
  - Izerskie Centrum Pulmonologii i Chemioterapii "Izer-Med" Sp. z o.o, Szklarska Poręba
  - Specjalistyczny Szpital Onkologiczny NU-MED, Tomaszów Mazowiecki
  - Centralny Szpital Kliniczny MSWiA w Warszawie, Warsaw
  - Pfizer Polska, Warsaw
  - Wojewodzki Szpital Specjalistyczny we Wroclawiu, Wroclaw
  - Dolnośląskie Centrum Onkologii, Wroclaw

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Radecka B, Zurawski B, Lacko A, Grela-Wojewoda AA, Wieruszewska-Kowalczyk K, Senkus-Konefka E. Real-world treatment patterns of hormone receptor-positive and human epidermal growth factor receptor 2-negative advanced breast cancer. Contemp Oncol (Pozn). 2025;29(4):370-376. doi: 10.5114/wo.2025.156076. Epub 2025 Nov 11. PMID 41438813
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A5481177